CLINICAL TRIAL: NCT07179653
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of TVAX-008 Injection in Chronic Hepatitis B Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grand Theravac Life Sciences (Nanjing) Co., Ltd. (Industry)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Sichuan Provincial People's Hospital (Other); Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other); Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YDSWX(TVAX-008)-005(II)
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: HBV Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TVAX-008 (Experimental)
  Interventions: Drug: TVAX-008
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TVAX-008 — TVAX-008
  Arms: TVAX-008
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
The objective of this study was to evaluate the efficacy and safety of TVAX- 008 injection in a multicenter, randomized, double-blind, placebo-controlled, parallel-group phase II clinical trial in subjects with HBSAg levels of 0.05 to 100 IU/mL, including CHB patients previously treated with siRNA/ASO drugs and treatment-naive HBV infection.

ELIGIBILITY:
Inclusion Criteria:

- aged 18~65 ； Serum HBsAg positive ≥ 6 months； HBeAg negative；

Exclusion Criteria:

* Treatment with interferon or pegylated interferon within 12 weeks prior to first use of investigational product; or planned treatment with interferon or pegylated interferon during the trial;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HBsAg clearance rate | Week49

CONTACTS AND LOCATIONS:
Locations (1):
- NanFang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided